CLINICAL TRIAL: NCT04288869
Title: Change in Brain Perfusion During Induction of General Anesthesia: Relationship Between Transcranial Doppler, Bispectral Index and Cerebral Oximetry : a Prospective Observational Study CERVO2
Brief Title: Change in Brain Perfusion During Induction of General Anesthesia
Acronym: CERVO2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: INSERM UMR-942, Paris, France (Other); LMS Ecole polytechnique (Unknown); M3DISIM Inria Université Paris-Saclay (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP190945; 2019-A02516-51 (Other: IDRCB)
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Interventional Radiology; Orthopedic Surgery
Keywords: cerebral perfusion; general anesthesia; hypotension; transcranial Doppler; Bispectral Index; Near-infrared spectroscopy
MeSH Terms: conditions — Hypotension | interventions — Ultrasonography, Doppler, Transcranial; Consciousness Monitors; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional radiology or surgery under general anesthesia: Monitoring of patients (mean arterial blood pressure, Transcranial Doppler , bispectral index, near infrared spectroscopy) who benefit from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anaesthesia during the interventional neuroradiology or orthopedic surgery in adults .
  Interventions: Other: Continuous monitoring of arterial blood pressure; Other: Transcranial Doppler; Other: Bispectral Index (BIS); Other: Near-infrared spectroscopy

INTERVENTIONS:
Other: Continuous monitoring of arterial blood pressure — For all patients, mean arterial pressure (unit mmHg) will be collected over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation.
Other: Transcranial Doppler — Measurement of cerebral blood flow velocity (CFV) with use of Transcranial Doppler ultrasonography.
  For all patients, CFV (unit cm/s) will be collected over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation.
Other: Bispectral Index (BIS) — Continuous measurement of burst suppression (BS; %) with use of Bispectral Index (BIS).
  For all patients, BS will be collected over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation
Other: Near-infrared spectroscopy — Continuous measurement of cerebral oxygen saturation (SO2) with Near-infrared spectroscopy (NIRS).
  For all patients, SO2 (%) will be collected over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation.

SUMMARY:
Arterial hypotension during general anesthesia remains a factor of poor outcomes, increases the risk of myocardial infarction, acute kidney injury and 1-year mortality. Furthermore, arterial hypotension may also decrease cerebral perfusion contributing to worsen neurological outcome. It seems necessary to monitor cerebral perfusion during anesthesia and to define individual dynamic targets of blood pressure. The goal of this study is to evaluate cerebral perfusion change in adult patients with or without cardiovascular risk factors during a standardized propofol-remifentanil anesthesia induction. Cerebral perfusion will be evaluated and compared by simultaneous measurements of cerebral blood flow, cerebral oxygen saturation and neurological function with use of transcranial Doppler (TCD), Near infrared spectroscopy (NIRS) and the Bispectral index (BIS) monitoring, respectively. Those measurements will be also repeated during and after treatment of arterial hypotension episodes in both groups.

DETAILED DESCRIPTION:
Main objective: blood pressure target to maintain cerebral perfusion is related to patient's characteristics or comorbidities, it remains uncertain which threshold of blood pressure is to use during general anesthesia in each specific case. Thus, it seems necessary to monitor the cerebral perfusion during anesthesia and to determine the individual dynamic targets of blood pressure. The measure of middle cerebral artery blood flow velocity by transcranial doppler (TCD) is a clinical method to assess cerebral perfusion during general anesthesia and several studies have reported the hemodynamic impact on cerebral blood flow during induction.

Cerebral perfusion can also be approached by near infrared spectroscopy (NIRS) which measures continuously cerebral oxygen saturation. Bispectral index (BIS), which allows a simplified form of continuous electroencephalogram monitoring to assess depth of anesthesia, could also provide the cerebral hypoperfusion assessment quantified by the count of burst suppression ratio (SR). Potentially, those tools need to be combined to assess cerebral perfusion properly.

The goal of this study is to evaluate cerebral perfusion change in adult participants with or without cardiovascular risk factors during a standardized propofol-remifentanil anesthesia induction. Cerebral perfusion will be evaluated and compared using simultaneously the TCD, NIRS and BIS measurements. Those measurements will be also repeated during and after treatment of arterial hypotension episodes in both groups.

Population concerned : the study involves major patients who benefit from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anesthesia during an interventional neuroradiology procedure or orthopedic surgery.

Research Proceedings: all monitoring (TCD, BIS, NIRS) will be collected from the healthy side, contralateral to the interventional side. BIS, NIRS and continuous non-invasive blood pressure measurement will be all connected to the main monitor. For all participants, the data from TCD, NIRS, BIS and the hemodynamic data will be collected over three distinct periods of the interventional procedure : (1) baseline or during preoxygenation at FiO2 of 21% (fraction of inspired oxygen) in awake patients, (2) before Orotracheal Intubation and (3) just after mechanical ventilation.

In patients presenting a hypotensive episode at any time of the procedure, all parameters will be collected before and at the peak effect after a 10μg bolus injection of norepinephrine.

Patients will be assigned to one of two groups according to the presence of cardiovascular risk factors. Major risk factor is age > 50 years old. Minor risk factors include history of congestive heart failure, history of cardiovascular event, current smoking, diabetes mellitus, dyslipidemia, arterial hypertension. Patients will be classified into the high-risk group (Hi-risk) if they have at least one major cardiovascular risk factor or two minor factors, or into the low risk group (Lo-risk) if they present one minor or no risk factors.

During their interventional neuroradiology procedure or orthopedic surgery, all patients' routine monitoring will consist in collecting the following parameters: electrocardiogram, pulsated oxygen saturation, endtidal CO2, respiratory rate, tidal volume and neuromuscular function.

For all patients whatever the comorbidities, anesthesia induction will be performed using a target-controlled infusion (Orchestra® Base Primea - Fresenius Kabi France). According to our standard of care, intra-operative episodes of hypotension (mean arterial pressure (MAP) < 65 mmHg or < 80% baseline) will be treated by Norepinephrine bolus of 10 μg.

Statistics: Changes in parameters across the time, during induction and/or during vasopressors boluses will be tested by using a paired Student-t test after testing the normality of the distribution. Correlation between the change in MAP and Vm during induction will be done using Spearman test. Complete analysis will also be performed to compare the Low-risk and High-risk patients. The analysis of vasopressor boluses will be performed depending on the time of administration: boluses which are given immediately after induction of anesthesia (early) and boluses given after a 30 minutes period of constant intravenous calculated concentrations of anesthesia (late). All statistical analyses will be performed using R statistical software (The 'R' Foundation for Statistical Computing, Vienna, Austria). Results will be expressed as means (± SD). A two sided p value of 0.05 will be considered significant.

The sample size calculation is based on the following assumptions: incidence of Hi-risk patients of 50%, as previously reported; incidence of burst suppression during induction in low risk patients of 20%; difference of incidence of burst suppression between low- and high-risk patients of 30%; power at 80% and type I error at 5%. Accordingly, the calculated sample size is 101 patients for the entire population.

ELIGIBILITY:
Inclusion Criteria:

* Major patients (≥ 18 years old)
* Eligible for an interventional radiology procedure or orthopedic surgery under general anesthesia.
* Patients who expressed their non-opposition to participation in this research

Exclusion Criteria:

* Patients under the age of 18.
* Patient opposed to participation in the protocol
* Pregnant woman
* Patient under judicial protection measure
* Patient without affiliation to a social security scheme-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study involves major patients who benefit from intraoperative hemodynamic optimization with norepinephrine (as noradrenaline tartrate) for maintaining blood pressure under general anesthesia during an interventional neuroradiology procedure or orthopedic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial blood pressure | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, the mean arterial pressure (unit mmHg) will be collected continuously, over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation
Cerebral blood flow velocity | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, CFV (unit cm/s) will be collected continuously, using Transcranial Doppler, over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation.
Burst Suppression | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  Continuous measurement of burst suppression (BS; %) with use of Bispectral Index (BIS) over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation.
Cerebral oxygen saturation | Duration of the surgical intervention or interventional neuroradiology procedure (maximum 1 day)
  For all patients, the cerebral oxygen saturation (SO2; %) will be collected continuously, using Near-infrared spectroscopy, over three distinct periods: 1) baseline or during pre-oxygenation at FiO2 of 21% in awake patients, 2) before orotracheal intubation, and 3) just after mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim MATEO, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Fabrice VALLEE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Lariboisière Hospital, Department of Anesthesiology and Intensive Care, Paris, France